CLINICAL TRIAL: NCT01679002
Title: Steady-state Pharmacokinetics of BIA 2-093 and Oxcarbazepine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-110
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Oxcarbazepine; Eslicarbazepine Acetate; BIA 2-093
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): BIA 2-093 900 mg once-daily period followed by BIA 2-093 450 mg twice-daily period followed by oxcarbazepine 450 mg twice-daily period
  BIA 2-093 450 mg od - BIA 2-093 450 mg bid - OXC 900 mg bid
  Interventions: Drug: BIA 2-093; Drug: Oxcarbazepine
- Group B (Experimental): BIA 2-093 450 mg twice-daily period followed by oxcarbazepine 450 mg twice-daily period followed by BIA 2-093 900 mg once-daily period
  BIA 2-093 450 mg bid - OXC 450 mg bid - BIA 2-093 900 mg od
  Interventions: Drug: BIA 2-093; Drug: Oxcarbazepine
- Group C (Experimental): oxcarbazepine 450 mg twice-daily period followed by BIA 2-093 900 mg once-daily period followed by BIA 2-093 450 mg twice-daily period
  OXC 450 mg bid - BIA 2-093 900 mg od - BIA 2-093 450 mg bid
  Interventions: Drug: BIA 2-093; Drug: Oxcarbazepine

INTERVENTIONS:
Drug: BIA 2-093
  Other Names: ESL, Eslicarbazepine acetate
Drug: Oxcarbazepine
  Other Names: OXC, Trileptal®

SUMMARY:
To investigate the steady-state pharmacokinetics of once-daily and twice-daily regimens of BIA 2-093 and twice-daily regimen of Oxcarbazepine (Trileptal®) in healthy subjects and to assess the tolerability of such regimens in healthy subjects.

DETAILED DESCRIPTION:
Single centre, open-label, randomised, three-way crossover study in 12 healthy volunteers. The study consisted of three 8-day treatment periods separated by washout periods of 10-15 days. On each of the treatment periods the volunteers received either a daily oral dose of BIA 2-093 900 mg once-daily (od), BIA 2-093 450 mg twice-daily (bid), or Oxcarbazepine (Trileptal®) 450 mg bid.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were eligible for entry into the study if they fulfilled the following inclusion criteria:
* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 28 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, neurological examination, and 12-lead ECG.
* Subjects who had clinical laboratory tests clinically acceptable.
* Subjects who were negative for HBsAg, anti-HCV Ab and HIV-1 and HIV-2 Ab tests at screening.
* Subjects who were negative for alcohol and drugs of abuse at screening and first admission.
* Subjects who were non-smokers or who smoked less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* If case of female subjects, subjects who were not of childbearing potential by reason of surgery or, if of childbearing potential, who used one of the following methods of contraception: double-barrier, intrauterine device or abstinence.
* If case of female subjects, subjects who had a negative pregnancy test at screening and first admission.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria.
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of hypersensitivity to carbamazepine or oxcarbazepine or any other relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 14 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening and/or first admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or first admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used prescription or over-the-counter medication within two weeks of first admission.
* Subjects who had used any investigational drug and/or participated in any clinical trial within four months of their first admission.
* Subjects who had previously received BIA 2-093.
* Subjects who had donated and/or received any blood or blood products within the previous 4 months prior to screening.
* Subjects who were vegetarians, vegans and/or have medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* In case of female subjects, subjects who were pregnant or breast-feeding.
* In case of female subjects, subjects who were of childbearing potential and did not use an approved effective contraceptive method or used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2003-10; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Vaz-da-Silva, MD, PhD, Principal Investigator — BIAL - Portela & Cª S.A.
Locations (1):
- BIAL - Portela & Cª S.A. - Human Pharmacology Unit (UFH), S. Mamede Do Coronado, Trofa, Portugal

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: BIA 2-093 900 mg once-daily period followed by BIA 2-093 450 mg twice-daily period followed by oxcarbazepine 450 mg twice-daily period.
  BIA 2-093 900 mg od - BIA 2-093 450 mg bid - OXC 450 mg bid
- Group B: BIA 2-093 450 mg twice-daily period followed by oxcarbazepine 450 mg twice-daily period followed by BIA 2-093 900 mg once-daily period
  BIA 2-093 450 mg bid OXC 450 mg bid BIA 2-093 900 mg od
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 4 | 4 | 4
BIA 2-093 900 mg Once-daily Period | 4 | 3 | 4
BIA 2-093 450 mg Twice-daily Period | 4 | 4 | 4
Oxcarbazepine 450 mg Twice-daily Period | 3 | 4 | 4
Completed | 3 | 3 | 4
Not Completed | 1 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: BIA 2-093 450 mg once-daily period followed by BIA 2-093 450 mg twice-daily period followed by oxcarbazepine 450 mg twice-daily period BIA 2-093 450 mg od - BIA 2-093 450 mg bid - OXC 450 mg bid
- Group B: BIA 2-093 450 mg twice-daily period followed by oxcarbazepine 450 mg twice-daily period followed by BIA 2-093 450 mg once-daily period BIA 2-093 450 mg bid - OXC 450 mg bid - BIA 2-093 450 mg od
- Group C: oxcarbazepine 450 mg twice-daily period followed by BIA 2-093 450 mg once-daily period followed by BIA 2-093 450 mg twice-daily period OXC 450 mg bid - BIA 2-093 450 mg od - BIA 2-093 450 mg bid
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 12
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Drug Concentration
Description: Cmax - maximum observed plasma drug concentration for BIA 2-093 metabolites:
  BIA 2-194 BIA 2-195 Oxcarbazepine
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72 and 96 h post-dose
Population: The results are related to overall population in the study devided by period of treatment.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 2-093 900 mg od: ESL, Eslicarbazepine acetate BIA 2-093 900 mg od
- BIA 2-093 450 mg Bid: ESL, Eslicarbazepine acetate BIA 2-093 450 mg bid
- Oxcarbazepine 450 mg Bid: OXC, Oxcarbazepine 450 mg bid
Arm/Group | BIA 2-093 900 mg od | BIA 2-093 450 mg Bid | Oxcarbazepine 450 mg Bid
Number analyzed (Participants) | 11 | 11 | 11
ng/mL
  Cmax (BIA 2-194) | 22210 (7257) | 16667 (3981) | 12195 (2053)
  Cmax (BIA 2-195) | 685 (188) | 702 (182) | 2481 (362)
  Cmax (Oxcarbazepine) | 208 (53.2) | 182 (47.2) | 1080 (548)

2. Secondary Outcome: AUC - Area Under the Plasma Concentration Versus Time Curve
Description: AUC - Area Under the Plasma Concentration Versus Time Curve for BIA 2-093 metabolites:
  BIA 2-194 BIA 2-195 Oxcarbazepine
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72 and 96 h post-dose
Population: The results are related to overall population in the study devided by period of treatment.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | BIA 2-093 900 mg od | BIA 2-093 450 mg Bid | Oxcarbazepine 450 mg Bid
Number analyzed (Participants) | 11 | 11 | 11
ng*h/mL
  AUC0-t (BIA 2-194) | 381601 (95368) | 283014 (74203) | 268376 (43294)
  AUC0-t (BIA 2-195) | 20164 (6790) | 19091 (6042) | 48841 (9041)
  AUC0-t (Oxcarbazepine) | 3238 (1033) | 2699 (909) | 5196 (1472)

3. Secondary Outcome: Number of of Subjects Reporting at Least One Adverse Event
Description: Number of of subjects reporting at least one adverse event.
Time Frame: 8 weeks
Population: The results are related to overall population in the study devided by period of treatment.
Measure: Number; unit: Subjects
Arm/Group | BIA 2-093 900 mg od | BIA 2-093 450 mg Bid | Oxcarbazepine 450 mg Bid
Number analyzed (Participants) | 11 | 12 | 11
Subjects | 9 | 10 | 11

ADVERSE EVENTS:
Groups:
- BIA 2-093 900 mg: ESL, Eslicarbazepine acetate BIA 2-093 900 mg od
Arm/Group | BIA 2-093 900 mg | BIA 2-093 450 mg Bid | Oxcarbazepine 450 mg Bid
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 9/11 | 10/12 | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 2-093 900 mg (N=11) | BIA 2-093 450 mg Bid (N=12) | Oxcarbazepine 450 mg Bid (N=11)
Asthenia (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1
Appetite lost (Metabolism and nutrition disorders) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Erection increased (Reproductive system and breast disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Blepharospasm (Eye disorders) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Increased libido (Psychiatric disorders) | 0 | 0 | 1
Diffuse macular rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 3 | 3 | 6
Dizziness (Nervous system disorders) | 0 | 2 | 6
Frontal headache (Nervous system disorders) | 2 | 1 | 2
Headache (Nervous system disorders) | 1 | 1 | 1
Nystagmus (Nervous system disorders) | 2 | 0 | 1
Orthostatic dizziness (Nervous system disorders) | 1 | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1
Concentration impairment (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Motor dysfunction NOS (Nervous system disorders) | 0 | 1 | 0
Numbness of limbs (Nervous system disorders) | 0 | 0 | 1
Occipital headache (Nervous system disorders) | 0 | 0 | 1
Vasovagal reaction (Nervous system disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal colic (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Dry lips (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric pain (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Heartburn (Gastrointestinal disorders) | 0 | 1 | 0
Loose stools (Gastrointestinal disorders) | 0 | 0 | 1
Right upper quadrant pain (Gastrointestinal disorders) | 0 | 1 | 0
Tooth pain (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes